CLINICAL TRIAL: NCT05286762
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled, Multi-center, Fixed-dose, Parallel Group Efficacy and Safety in Pediatrics (6-17) With Attention-Deficit/Hyperactivity Disorder (ADHD) Using CTx-1301 (Dexmethylphenidate)
Brief Title: Phase 3 Efficacy and Safety Fixed-Dose Study in Pediatrics (6-17) With ADHD Using CTx-1301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cingulate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTx-1301-005
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder; ADHD - Combined Type; Attention Deficit Hyperactivity Disorder Combined; Attention-deficit Hyperactivity; Attention Deficit Hyper Activity
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Random Allocation

STUDY DESIGN:
Intervention Model Description: Subjects are randomized in 1:1:1:1 order
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 18.75 mg CTx-1301 (dexmethylphenidate tablet) (Active Comparator): Subjects who are randomized to active drug (18.75 mg of CTx-1301) will be titrated (increased) weekly up to their assigned fixed dose. The starting dose at Day 0 is 12.5 mg; at week 1 they will be increased to their assigned dose of 18.75 mg. Subjects will remain on this assigned fixed dose for the remainder of the randomized study period.
  Interventions: Drug: CTx-1301-Dexmethylphenidate 12.5 mg (titration only); Drug: CTx-1301-Dexmethylphenidate 18.75mg (randomized fixed dose)
- 25 mg CTx-1301 (dexmethylphenidate tablet) (Active Comparator): Subjects who are randomized to active drug (25 mg of CTx-1301) will be titrated (increased) weekly up to their assigned fixed dose. The starting dose at Day 0 is 12.5 mg; at week 1 they will be increased to 18.75 mg; at week 2 they will be increased to their assigned dose of 25 mg. Subjects will remain on this assigned fixed dose for the remainder of the randomized study period.
  Interventions: Drug: CTx-1301-Dexmethylphenidate 12.5 mg (titration only); Drug: CTx-1301-Dexmethylphenidate 18.75mg (randomized fixed dose); Drug: CTx-1301-Dexmethylphenidate 25mg (randomized fixed dose)
- 37.5 mg CTx-1301 (dexmethylphenidate tablet) (Active Comparator): Subjects who are randomized to active drug (37.5 mg of CTx-1301) will be titrated (increased) weekly up to their assigned fixed dose. The starting dose at Day 0 is 12.5 mg; at week 1 they will be increased to 18.75 mg; at week 2 they will be increased to 25 mg; at week 3 they will be increased to their assigned dose of 37.5 mg. Subjects will remain on this assigned fixed dose for the remainder of the randomized study period.
  Interventions: Drug: CTx-1301-Dexmethylphenidate 12.5 mg (titration only); Drug: CTx-1301-Dexmethylphenidate 18.75mg (randomized fixed dose); Drug: CTx-1301-Dexmethylphenidate 25mg (randomized fixed dose); Drug: CTx-1301-Dexmethylphenidate 37.5 mg (randomized fixed dose)
- Placebo (Placebo Comparator): Subjects randomized to placebo will be on placebo for the full 5 weeks of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CTx-1301-Dexmethylphenidate 12.5 mg (titration only) — Subjects will be randomized at Visit 2 to CTx-1301 to 12.5mg
  Other Names: d-MPH
  Arms: 18.75 mg CTx-1301 (dexmethylphenidate tablet); 25 mg CTx-1301 (dexmethylphenidate tablet); 37.5 mg CTx-1301 (dexmethylphenidate tablet)
Drug: CTx-1301-Dexmethylphenidate 18.75mg (randomized fixed dose) — Subjects will be randomized at Visit 2 to CTx-1301 to 12.5mg, then week 1 to 18.75 mg
  Other Names: d-MPH
  Arms: 18.75 mg CTx-1301 (dexmethylphenidate tablet); 25 mg CTx-1301 (dexmethylphenidate tablet); 37.5 mg CTx-1301 (dexmethylphenidate tablet)
Drug: CTx-1301-Dexmethylphenidate 25mg (randomized fixed dose) — Subjects will be randomized at Visit 2 to CTx-1301 to 12.5mg, then week 1 to 18.75 mg, then week 2 to 25 mg
  Other Names: d-MPH
  Arms: 25 mg CTx-1301 (dexmethylphenidate tablet); 37.5 mg CTx-1301 (dexmethylphenidate tablet)
Drug: CTx-1301-Dexmethylphenidate 37.5 mg (randomized fixed dose) — Subjects will be randomized at Visit 2 to CTx-1301 to 12.5mg, then week 1 to 18.75 mg, then week 2 to 25 mg, then week 3 to 37.5 mg
  Other Names: d-MPH
  Arms: 37.5 mg CTx-1301 (dexmethylphenidate tablet)
Drug: Placebo — Subjects will be randomized at Visit 2 to Placebo
  Arms: Placebo

SUMMARY:
A Phase 3, randomized, double-blind, placebo-controlled, multi-center, fixed-dose, parallel-group efficacy and safety study in a pediatric population (6-17) with Attention-Deficit/Hyperactivity Disorder (ADHD) using CTx-1301 (d-MPH). The study will be comprised of a screening period, a double-blind randomized phase, and a safety follow-up visit.

DETAILED DESCRIPTION:
A Phase 3, double-blind, randomized, placebo-controlled, multi-center, fixed-dose, parallel group efficacy and safety study in pediatrics (6-17) with ADHD diagnosis confirmed by an ADHD-RS-5 score of at least 28 and CGI-S score of at least 4 (moderately ill) at screening. The study will be comprised of a screening period, a double-blind randomized phase, and a safety follow-up visit.

The Study will be comprised of 3 periods:

* Screening Period (Day -30 to Day -1): Subjects will undergo a Screening Visit (Visit 1) up to 30 days prior to entering the randomized treatment period. Only subjects that meet all inclusion and no exclusion criteria at screening may be considered for entry/randomization into the study. A reminder telephone call will be completed 5 days prior to Day 0 (Visit 2) to ensure washout of current prohibited medications, to confirm inclusion/exclusion criteria, and to confirm date of next visit.
* Randomized Treatment Period (Day 0 to Day 35 +/- 3 days): Subjects will be randomized on Day 0 to active or placebo (placebo, CTx-1301 18.75 mg, CTx-1301 25 mg, or CTx-1301 37.5 mg). Subjects randomized to the active dose will have a starting dose of 12.5 mg on Day 0. Each subject randomized to an active dose will be titrated (increased) weekly until they reach their assigned fixed dose; subjects must be on their assigned fixed dose a minimum of 2 sequential weeks prior to the primary efficacy assessment at Week 5/Visit 8. Subjects will be instructed to take their dose every morning at-home upon waking, no later than 8:00 am.
* Safety Follow-Up Visit (Day 42 +/- 5 days): Subjects will be evaluated for safety after washout of medication.

Subjects will participate in the study as outpatients for up to approximately 10 weeks (including screening); a 30-day screening period, a 5-week double-blind randomized period, and a 1-week follow-up safety visit.

Completion of the primary study is defined as LSLV at Visit 9.

Subjects will be randomized at baseline to CTx-1301 or placebo (CTx-1301 18.75 mg, CTx-1301 25 mg, CTx-1301 37.5 mg, or placebo). Starting dose for subjects randomized to active treatment is 12.5 mg. These subjects will then be titrated up to their assigned fixed dose (18.75, 25, or 37.5 mg) for the last two weeks of the study period. Subjects randomized to placebo will receive placebo treatment for the full 5 weeks of the study.

Sparse PK sampling will be conducted after a single dose and at steady state from the patient population with special attention given to the time the sample is obtained post-dose. These analyses will inform strategies that manage dosing and detail administration for a given subpopulation, planned subsequent studies, and support labeling.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 6 and 17 years of age (inclusive) at the time of Randomization (Visit 2). Subjects who are expected to turn 18 years of age during the trial will not be allowed.
2. Subject must have a body weight between the 5th and 95th percentile (≥5th percentile and ≤95th percentile) for their respective age and sex.
3. Subject is unsatisfied with his/her current pharmacological therapy for treatment of ADHD or not currently receiving pharmacological therapy for ADHD. Inclusion of subjects who are naïve to pharmacological therapy for ADHD is permitted.
4. Subjects of child-bearing potential at screening or that become of child-bearing potential during the study must agree to remain abstinent or agree to use a highly effective, medically acceptable form of birth control for the time of written assent and for at least 30 days after the last dose of study drug has been taken (females). Male subjects with female partners must agree at Screening to remain abstinent or agree to use an effective and medically acceptable form of birth control from Screening to 90 days after the last dose of study drug. Child-bearing potential is defined as any female who has had their first period or is 12 years or older (or will be 12 while in the study).
5. Subject must be in general good health defined as absence of any clinically relevant abnormalities as determined by the Investigator based on physical and neurological examinations, vital signs, ECGs (QTc less than or equal to 460 milliseconds), medical history, and laboratory values (hematology, chemistry, serology, TSH, or urinalysis) at Screening. If any of the exams or values are not within the laboratory reference range, the Investigator must review range and determine if clinically relevant. If clinically relevant, the subject is not eligible for the study.
6. Subject's intellectual function is at an age-appropriate level, as deemed by the Investigator.
7. Subject must meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for the primary diagnosis of ADHD or any of the three presentations (combined, inattentive, or hyperactive/impulsive presentation) upon clinical evaluation and confirmed by the MINI International Neuropsychiatric Interview of Children and Adolescents (MINI-KID). The MINI should also be used to evaluate any other psychotic disorders.
8. Subject must score 28 or higher on the ADHD-RS-5 scale at the Baseline visit (Visit 2).
9. Subject must have a score of 4 (moderately ill) or higher on the clinician-administrated Clinical Global Impressions-Severity (CGI-S) scale at Baseline (Visit 2).
10. Subject must be able and willing to wash out of stimulant ADHD medications (except study drug as indicated per protocol), including herbal medication, from 5 days prior to the start of the randomized phase (Visit 2) and for the duration of the entire study, defined as completion of the safety follow-up visit (approximately 1.25 months, excluding screening). Additionally, subject must be able and willing to wash out from non-stimulant ADHD medications 21 days prior to the start of the randomized phase (Visit 2) and for the duration of the entire study (approximately 1.25 months, excluding screening), defined as completion of the safety follow-up visit.
11. Subject and parent/legal guardian, and/or caregiver (if applicable) must be able to read, write, speak, and understand English and be able to communicate with the Investigator and study coordinator in a satisfactory fashion and complete any study-related materials. Subject and parent/legal guardian, and/or caregiver (if applicable) must plan to be available for the entire duration of the study.
12. One or more of the parents/legal guardians/caregivers of the subject must voluntarily give written permission for him/her to participate in the study.
13. Subject must provide written assent prior to study participation.
14. Subject, subject's parent/legal guardian, and/or caregiver (if applicable) must understand and be willing and able to comply with study procedures as well as the visit schedule. If the subject is cared for by a caregiver for relevant portions of the day, the caregiver may be more suitable for certain assessments, and the caregiver will need to agree to the applicable procedures and visits.
15. Subject must be able to swallow the CTx-1301 tablet as evidenced by ability to swallow a similar size tablet (placebo) at screening.

Exclusion Criteria:

1. If female and of child-bearing potential, the subject must not be pregnant or breastfeeding at any time during the study or for 30 days following the completion of the study, defined as completion of safety visit at the end of study (Visit 9). If of child-bearing potential, urine hCG tests will be administered at protocol-specified time points. Any positive pregnancy test during the study will exclude them from further participation in the study.
2. Subject has any psychiatric diagnosis of bipolar I or II disorder, major depressive disorder, conduct disorder, disruptive mood dysregulation disorder (DMDD), intellectual disability, obsessive-compulsive disorder, eating disorder, anxiety disorder (including generalized anxiety disorder), any history of psychosis, autism spectrum disorder, a history of motor or vocal tics or Tourette's Syndrome, confirmed genetic disorder with cognitive and/or behavioral disturbances, or any other diagnosis/significant medical history that at the discretion of the Investigator excludes the subject from entry into the study.
3. Subject has evidence of any chronic disease of the central nervous system (CNS) such as tumors, inflammation, seizure disorder, vascular disorder, potential CNS-related disorders that might occur in childhood, or history of persistent neurological symptoms related to a serious head injury.
4. Subject has any clinically significant and/or unstable/uncontrolled medical abnormality or chronic medical condition, persistent neurological symptoms, history of cardiovascular abnormality, abnormalities of respiratory, hepatic, gastrointestinal, renal, or any disorder or history of a condition that would impact or interfere with drug absorption, distribution, metabolism, or excretion during the study or may interfere with the participants ability to participate in the study.
5. Subject has family history of early cardiovascular disease or sudden death.
6. Subject has any history of attempted suicide or clinically significant suicidal ideation based on the Columbia Suicide Severity Rating Scale (C-SSRS) assessment, or answers "yes" to "Suicidal Ideation" item 4 or 5 of any lifetime history on the C-SSRS Children's Lifetime/Recent assessment at screening.
7. Subject has history of seizures, excluding febrile seizures.
8. Subject has a known primary sleep disorder (e.g., sleep apnea, narcolepsy, etc.)
9. If the subject's blood pressure is < 90th percentile for their age, sex, and height, the single read is sufficient. If the subject's blood pressure is ≥ 90th percentile, two additional reads will be taken, and the three reads will be averaged. If the average of the three readings is ≥ 95th percentile at screening they will be excluded.
10. Subject is considered treatment refractory by the Investigator or is intolerant to stimulant ADHD mediation.
11. Any use of anticonvulsants currently or within the past 2 years.
12. Uncontrolled thyroid disorder indicated by thyroid stimulating hormone (TSH) ≤0.8 x the lower limit of normal (LLN) or ≥ 1.25 x the upper limit of normal (ULN) from the reference laboratory.
13. Subject has first-degree relatives (biological parent or sibling) with a history of schizophrenia, schizoaffective disorder, bipolar I disorder, or bipolar II disorder.
14. Subject has history of substance abuse or shows evidence of substance use or has a positive urine drug screen at Screening or Baseline. Subjects with positive drug screens may be allowed to continue in the study if the result of the positive drug screen is from prescribed medications and the subject is willing to washout of the medication as required per protocol.
15. Previous treatment experience/exposure to CTx-1301.
16. Subject has a history of allergic reaction or sensitivity to methylphenidate, dexmethylphenidate, or any other substance contained in CTx-1301 or the placebo drug.
17. Subject has participated in any other clinical study with an investigational drug/product within 30 days prior to Screening or is currently participating in another clinical study.
18. Subject's family anticipates a move outside the geographic range of the investigative site during the duration of the study period or plans on travel that would not allow compliance to the protocol during the study period.
19. Subject is unsuitable in any other way, to participate in the study, as determined by the Investigator.
20. Subject is a family member of an employee at the study center, of the investigator, or those with direct involvement in the proposed study under the direction of that investigator or study center.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Based on gender as defined at birth.
Enrollment: 103 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Brams, MD, Study Director — Cingulate; Ann Childress, MD, Study Chair — Center for Psychiatry And Behavioral Medicine Inc.
Locations (24):
- United States (24):
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Meridien Research, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Sisu Bhr, Llc, Springfield, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - St Charles Psychiatric Associates & Midwest Research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine. Inc., Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Dayton Clinical Research, Dayton, Ohio
  - SP Research PLLC, Oklahoma City, Oklahoma
  - Summit Research Network, LLC, Portland, Oregon
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Access Clinical Trials Inc., Nashville, Tennessee
  - BioBehavioral Research of Austin, Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - Houston Clinical Trials, Bellaire, Texas
  - FutureSearch Trials, Dallas, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Family Psychiatry of The Woodlands, Woodland, Texas
  - Clinical Research Partners LLC, Petersburg, Virginia

IPD SHARING:
Plan to Share IPD: No
Overall study data as required by FDAAA801 will be shared upon completion of the study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Although approximately 385 subjects were expected to enroll in the study, the study was completed with 103 subjects enrolled after an agreement was reached with FDA on the requirements necessary for filing an NDA for CTx-1301. Subjects were recruited at 24 sites from August 1, 2023 to December 13, 2023.
Pre-assignment Details: Of the 168 screened subjects, 103 subjects were randomized and received treatment in the study, with a similar number of subjects in each treatment group.
Period: Overall Study
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Started | 26 | 26 | 25 | 26
Completed | 21 | 24 | 21 | 22
Not Completed | 5 | 2 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 25 | 26 | 103
Age, Customized [Count of Participants; unit: Participants]
  6-12 Years | 16 | 16 | 16 | 16 | 64
  13-17 Years | 10 | 10 | 9 | 10 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 9 | 9 | 41
  Male | 13 | 16 | 16 | 17 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 4 | 6 | 19
  Not Hispanic or Latino | 20 | 23 | 21 | 20 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 12 | 14 | 13 | 51
  White | 11 | 11 | 11 | 12 | 45
  More than one race | 3 | 2 | 0 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 25 | 26 | 103
BMI Z-Score [Mean (Standard Deviation); unit: Z-Score] — BMI Z-scores were calculated using the CDC source code SAS program. BMI z-scores for children measure how a child's BMI compares to to other children of the same age and sex, indicating if they are underweight, healthy, overweight, or obese based on standard deviations (SD) from the average (z-score of 0). Positive scores are above average (greater than or equal to 1 SD for overweight, greater than or equal to 2 SD for obesity), and negative scores are below average (less than or equal to -2 SD for thinness).
  Z-Score | 0.413 (0.8340) | 0.221 (1.0205) | 0.314 (1.1993) | 0.315 (0.9324) | 0.315 (0.9909)
BMI Percentile [Mean (Standard Deviation); unit: Percentile] — BMI percentiles were calculated using the CDC source code SAS program.
  Percentile | 62.84 (27.212) | 56.31 (31.410) | 62.40 (31.393) | 60.18 (29.309) | 60.41 (29.538)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Analysis Will Analyze the Mean Change From Baseline (Pre-dose) at Visit 2 of Attention Deficit Hyperactivity Disorder Rating Scale 5 (ADHD-RS-5) Scores to ADHD-RS-5 at Visit 8.
Description: The Attention Deficit Hyperactivity Disorder Rating Scale Version 5 (ADHD-RS-5) overall scores range from 0-54; an improvement from Baseline is defined as a decrease in the overall score.
Time Frame: Baseline (Day 0) to Week 5 (Visit 8)
Population: Summary of observed values and changes from Baseline to Week 5 in the ADHD-RS-5 total score for all subjects (Intent-to-Treat Set).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 22
score on a scale | -18.0 (12.24) | -17.8 (12.78) | -22.0 (15.07) | -8.1 (13.88)

2. Secondary Outcome: The Primary Efficacy Analysis Will Analyze the Mean Change From Baseline (Pre-dose) at Visit 2 of Clinical Global Impression - Severity (CGI-S) Scores to CGI-S at Visit 8.
Description: The Clinical Global Impression - Severity (CGI-S) is a single score ranging from 1-7; an improvement from Baseline is defined as a decrease in the score.
Time Frame: Baseline (Day 0) to Week 5 (Visit 8)
Population: Summary of CGI-S score and change from Baseline to Week 5 for all subjects (Intent-to Treat Set)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Number analyzed (Participants) | 21 | 22 | 20 | 22
score on a scale | -1.5 (1.33) | -1.5 (1.22) | -2.2 (1.57) | -0.8 (1.34)

3. Secondary Outcome: Safety - Number of Subjects With Clinically Significant Changes in Vital Signs That Resulted in an Adverse Event.
Description: Vital signs will be evaluated in each in-office visit; clinically significant changes will be recorded as an adverse event.
Time Frame: Baseline to Visit 8 (5 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Number analyzed (Participants) | 26 | 26 | 25 | 26
Participants | 2 | 2 | 3 | 1

4. Secondary Outcome: Safety - Number of Subjects With Clinically Significant Changes in Blood Labs That Resulted in an Adverse Event.
Description: Safety labs will be taken at Screening to determine eligibility for entry into the study; safety labs are assessed again at Visit 8 and any clinically significant change from Screening labs will be recorded as an adverse event.
Time Frame: Screening to Visit 8 (approximately 5-9 weeks, depending on screening window)
Measure: Count of Participants; unit: Participants
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Number analyzed (Participants) | 26 | 26 | 25 | 26
Participants | 0 | 0 | 1 | 1

5. Secondary Outcome: Safety - Number of Subjects With Clinically Significant Changes in Physical Exam Findings That Resulted in an Adverse Event.
Description: Physical exams will be conducted at Screening, Baseline, and Visit 8. Changes noted as clinically significant from Baseline to Visit 8 will be recorded as an adverse event.
Time Frame: Baseline to Visit 8 (5 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Number analyzed (Participants) | 26 | 26 | 25 | 26
Participants | 11 | 14 | 17 | 8

6. Secondary Outcome: Safety - Number of Subjects With Clinically Significant Changes in Height and Weight BMI That Resulted in an Adverse Event.
Description: Height and Weight (BMI) will be evaluated at all in-office visits. Any clinically significant change in BMI from Baseline to Visit 8 will be recorded as an AE.
Time Frame: Baseline to Visit 8 (5 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Number analyzed (Participants) | 26 | 26 | 25 | 26
Participants | 0 | 0 | 2 | 0

7. Secondary Outcome: Safety - Number of Subjects With Clinically Significant Changes in C-SSRS Findings That Resulted in an Adverse Event.
Description: C-SSRS will be conducted at all in-office visits. Any clinically significant change from Baseline (at any visit) will be reported as an AE.
Time Frame: Baseline to Visit 8 (5 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Number analyzed (Participants) | 26 | 26 | 25 | 26
Participants | 0 | 0 | 1 | 0

8. Secondary Outcome: Safety - Number of Subjects With Clinically Significant Changes in ECG Findings That Resulted in an Adverse Event.
Description: ECGs will be taken at Screening to determine eligibility for entry into the study; ECGs are assessed again at Visit 8 and any clinically significant change from Screening ECG will be recorded as an adverse event.
Time Frame: Screening to Visit 8 (approximately 5-9 weeks, depending on screening window)
Measure: Count of Participants; unit: Participants
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Number analyzed (Participants) | 26 | 26 | 25 | 26
Participants | 1 | 2 | 1 | 1

9. Secondary Outcome: Safety - Incidence of TEAEs
Description: Treatment Emergent Adverse Events will be evaluated at each visit.
Time Frame: Screening to Visit 9 (approximately 6-10 weeks, depending on screening window)
Population: Overall summary of adverse events (Safety Set)
Measure: Count of Participants; unit: Participants
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
Number analyzed (Participants) | 26 | 26 | 25 | 26
Participants | 13 | 9 | 17 | 10

ADVERSE EVENTS:
Time Frame: Day -30 to Day 42
Arm/Group | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 13/26 | 9/26 | 17/25 | 10/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18.75 mg CTx-1301 (Dexmethylphenidate Tablet) (N=26) | 25 mg CTx-1301 (Dexmethylphenidate Tablet) (N=26) | 37.5 mg CTx-1301 (Dexmethylphenidate Tablet) (N=25) | Placebo (N=26)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 7 (7) | 0 (0)
Blood pressure increased (Investigations) | 1 (2) | 0 (0) | 2 (3) | 1 (1)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diastolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prehypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT05286762/Prot_SAP_000.pdf